CLINICAL TRIAL: NCT05634837
Title: Application of Clinical Decision Support System to Assist Pregnant Women to Increase Mediterranean Diet Adherence : A Randomised Controlled Trial
Brief Title: Increase in MedDiet Adherence in Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harokopio University (Other)
Collaborators: Iaso Maternity Hospital, Athens, Greece (Other)
Responsible Party: Principal Investigator, Andriana C Kaliora, Associate Professor, Harokopio University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PREGNANT_MEDDIET
Record Dates: First submitted 2022-11-08; First posted 2022-12-02 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Pregnancy Related

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Decision Support System counseling (Experimental): In the Intervention group (CDSS group), women receive a personalised daily dietary plan based on the Mediterranean diet and according to participant's needs, habits and preferences.
  Interventions: Behavioral: Decision Support System counseling
- Standard nutritional counseling (Other): Participants of the Control group did not have access to CDSS and only received general lifestyle guidelines.
  Interventions: Behavioral: Standard nutritional counseling

INTERVENTIONS:
Behavioral: Decision Support System counseling — Decision Support System counseling to improve diet and lifestyle in pregnancy
  Arms: Decision Support System counseling
Behavioral: Standard nutritional counseling — Counseling to improve diet and lifestyle in pregnancy
  Arms: Standard nutritional counseling

SUMMARY:
In the present randomised-controlled 3-month dietary intervention, we aim to a) increase Mediterranean diet adherence among apparently healthy pregnant women with the support of CDSS, and b) assess nutritional status and psychological parameters (anxiety and depression). To our knowledge, this is the first attempt investigating the effectiveness of CDSS in Mediterranean diet adherence of pregnant women.

DETAILED DESCRIPTION:
In this two-armed, single center, randomised controlled 3-month trial, apparently healthy pregnant women are randomly assigned to either the Control or the Intervention arm. The appointed statistician applies simple randomisation through a computer-generated randomization sequence. Treatment allocation is exposed to the statistician only after the assessment of outcomes.

At baseline before the start of the trial, each enrolled participant is appointed to a well-experienced dietician. In the Intervention group (CDSS group), women receive a personalised daily dietary plan based on the Mediterranean diet and according to participant's needs, habits and preferences. All elements needed for the synthesis of the dietary plan i.e., gestational age, body mass index (BMI) before the fetus conception, daily total energy expenditure, physical activity level based on the concept of metabolic equivalent of task (MET), caloric needs according to nutritional status, and macronutrient distribution are calculated using the CDSS database. The CDSS-dietary regimen consists of a daily eating program that was renewed every 15 days, paired with nutritional recommendations that are in line with the "National Dietary Guidelines for Pregnancy" [http://www.diatrofikoiodigoi.gr/?page=summary-women].

Before the start of the trial, women are trained to use the CDSS and receive individual login passwords. On a weekly basis, participants are instructed to input a 3-day food diary in the CDSS, made automatically available to the dieticians. When entering the CDSS, women monitor their personal goals i.e., body weight, physical activity, consumption of fruits and vegetables. Every other week, phone interviews are also performed to support nutritional and lifestyle consultation. Additionally, unexpected phone calls are made to obtain 24-hour dietary recalls.

Participants of the Control group do not have access to CDSS and only received general lifestyle guidelines based on the "National Dietary Guidelines for Pregnancy" via scheduled phone calls every 15 days with the appointed dietician. Women of the Control group are instructed to keep a 3-day food diary every week, sent by e-mail to the appointed dietician. Again, unexpected phone calls are made to obtain 24-hour dietary recalls.

ELIGIBILITY:
Inclusion Criteria:

* healthy pregnant women over 18 years

Exclusion Criteria:

* any metabolic disorder

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — pregnant women were eligible for the study
Enrollment: 40 (Actual)
Dates: Start 2019-05-31 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2023-01-13 (Actual)

PRIMARY OUTCOMES:
Change in the Mediterranean diet adherence | 3 months
  Differences in MedDiet adherence will be assessed by MedDiet score.

SECONDARY OUTCOMES:
Changes in anthropometric parameters | 3 months
  Changes in fat free mass (%) assessed by bioelectrical impedance
Changes in blood parameters | 3 months
  Changes in blood lipids measured in a biochemical analyzer
Changes in dietary intake | 3 months
  Changes in nutrient intake estimated by the nutritionist Pro analysis of 24h recalls
Changes in Hospital Anxiety and Depression Scale | 3 months
  Changes in well-being by applying a self-assessment scale (the Hospital Anxiety and Depression Scale) that comprises 14 items. Women with scores above 7 were at risk of having anxiety or depressive disorders

CONTACTS AND LOCATIONS:
Overall Officials: Andriana C. Kaliora, Study Director — HAROKOPIO UNIVERSITY OF ATHENS
Locations (1):
- Andriana Kaliora, Athens, Greece

IPD SHARING:
Plan to Share IPD: No